CLINICAL TRIAL: NCT03746782
Title: Investigating Synergistic Effects of Apixaban With Dual Anti-Platelet Therapy (DAPT) in Lowering Platelet Reactivity and Thrombin Generation
Brief Title: Apixaban + DAPT in Lowering Platelet Reactivity and Thrombin Generation
Acronym: SEARCH
Status: Completed | Type: Observational
Sponsor: CirQuest Labs, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: CV185-511 / CQ-15-10-005
Record Dates: First submitted 2018-07-11; First posted 2018-11-20 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Dual Anti-Platelet Therapy
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- ACS using clopidogrel + aspirin: Apixaban combined with blood specimens (in vitro) from Acute Coronary Syndrome participants prescribed a regimen of DAPT in the form of clopidogrel + aspirin
  Interventions: Diagnostic Test: Flow Cytrometry; Thrombin Generation Assay
- ACS using ticagrelor + aspirin: Apixaban combined with blood specimens (in vitro) from Acute Coronary Syndrome participants prescribed a regimen of DAPT in the form of ticagrelor + aspirin
  Interventions: Diagnostic Test: Flow Cytrometry; Thrombin Generation Assay
- Healthy Donors: Apixaban combined with blood specimens (in vitro) from healthy participants
  Interventions: Diagnostic Test: Flow Cytrometry; Thrombin Generation Assay

INTERVENTIONS:
Diagnostic Test: Flow Cytrometry; Thrombin Generation Assay — Apixaban combined with blood specimens (in vitro) of study participants

SUMMARY:
Investigating Synergistic Effects of Apixaban with Dual Anti-Platelet Therapy (DAPT) in Lowering Platelet Reactivity and Thrombin Generation

DETAILED DESCRIPTION:
Combination anti-platelet therapies particularly those combining aspirin with a P2Y12 antagonist (DAPT) are regarded as the current standard of care therapy for patients with Acute Coronary Syndrome (ACS). As thrombin potently induces platelet dense granular release and causes secondary adenosine 5'-diphosphate (ADP)-mediated P2Y12 receptor activation, apixaban via inhibition of thrombin generation may exhibit synergistic activity with direct P2Y12 receptor blockers such as clopidogrel or ticagrelor. The results from the study will provide a clearer understanding of how these antithrombotic agents work in combination and how the anti-Xa, apixaban, may reduce the contribution of thrombin and general platelet reactivity when used alone and in combination with antiplatelet agents. This study does NOT involve administration of medication to subjects. Experiments will be performed on donated blood samples from participants.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures (i.e., venipuncture).
2. Male or female at least 18 years of age but equal to or less than 75 years of age.
3. Females must be post-menopausal for at least one year or surgically sterile for at least 6 months.
4. For ACS Subjects:

   1. Documented prior history of ACS within the past 12 months.
   2. Currently prescribed a DAPT medication regimen of aspirin (81mg) plus a P2Y12 inhibitor, clopidogrel or ticagrelor, and none of the excluded medications listed in Exclusion Criteria #4.
   3. Have taken DAPT medication for at least 7 days as prescribed prior to blood collection.
5. For Healthy Subjects:

   1. Currently not prescribed and/or taking any of the excluded medications listed in Exclusion Criteria #4.

Exclusion Criteria:

1. Male or female less than 18 or greater than 75 years of age.
2. No prior history of ACS within 12 months (unless Healthy Subject)
3. Pregnancy
4. Currently prescribed and/or taking any of the following medications:

   Within the last 1 month:
   * PAR-1 antagonist (vorapaxar/Zontivity®)
   * Coumadin®
   * Heparin including low molecular weight heparin (enoxaparin/Lovenox®)
   * Factor Xa inhibitors (rivaroxaban/Xarelto®, apixaban/Eliquis®, edoxaban/Savaysa®, betrixaban/Bevyxxa®)
   * Direct thrombin inhibitors (hirudin, bivalirudin/Angiomax®, dabigatran/Pradaxa®)

   Within last 10 days:
   * Glycoprotein IIb/IIIa inhibitors (Eptifibatide/Integrilin®, Tirofiban/Aggrastat®, Abciximab/ReoPro®)
   * Acetylsalicylic Acid/Aspirin products (Alka-Seltzer®, Goody Powder®, BC Powder®, Pepto Bismol®, Aggrenox®) (except aspirin as prescribed for DAPT participants)

   Within last 3 days:
   * Phosphodiesterase inhibitors (cilostazol/Pletal®)
   * Adenosine reuptake inhibitors (dipyridamole/Persantine®)
   * NSAIDs
   * Decongestants
   * Antidepressants or Anti-anxiety medications:
   * Selective Serotonin Reuptake Inhibitors (SSRI) (fluoxetine/Prozac®, sertraline/Zoloft®, paroxetine/Paxil®)
   * Selective Norepinephrine Reuptake Inhibitors (SNRI) (venlafaxine/Effexor® or duloxetine/Cymbalta®)
5. Diagnosed with or possessing significant renal dysfunction as defined by the physician/investigator.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 subjects with ACS diagnosis and dual anti-platelet therapy requirements and 10 healthy subjects; no restrictions on gender, race or ethnicity; ages 18-74, non-childbearing potential for females.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Synergistic effects of in-vitro apixaban | 1 day
  Synergistic effects of in-vitro apixaban with antiplatelet agents in inhibiting platelet reactivity and thrombin generation

CONTACTS AND LOCATIONS:
Locations (1):
- CirQuest Labs, LLC, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided